CLINICAL TRIAL: NCT06012461
Title: Safety and Effectiveness of Closed-loop DBS in Parkinson's Disease: A Long-term Follow-up Study
Brief Title: Closed-loop DBS in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tsinghua University (Other)
Collaborators: National Engineering Research Center of Neuromodulation, Tsinghua University (Unknown); Beijing Tiantan Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Luming Li, Professor, Tsinghua University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDBS_PD_2023
Record Dates: First submitted 2023-06-18; First posted 2023-08-25 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Deep Brain Stimulation; Closed-loop DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral STN DBS Modulation (Experimental): Participants will be implanted with bilateral STN DBS using PINS 106RS system. DBS stimulation will be initiated one month post surgery. Follow-up visits will be conducted 1/3/6/9/12/15 months post surgery with clinical evaluation, STN LFP recording and resting state functional MRI testing. During the 6-15 month's visit, short-term closed-loop DBS modulation (from 24hours to 72hours ) will be conducted to test the safety and efficacy of closed-loop DBS therapy.
  Interventions: Other: Closed-loop DBS stimulation for 24 hours; Other: Open-loop DBS stimulation for 24 hours; Other: Closed-loop DBS stimulation for 72 hours; Other: Open-loop DBS stimulation for 72 hours

INTERVENTIONS:
Other: Closed-loop DBS stimulation for 24 hours — Continuous closed-loop modulation for 24 hours
Other: Open-loop DBS stimulation for 24 hours — Continuous open-loop modulation for 24 hours
Other: Closed-loop DBS stimulation for 72 hours — Continuous closed-loop modulation for 72 hours
Other: Open-loop DBS stimulation for 72 hours — Continuous open-loop modulation for 72 hours

SUMMARY:
Closed-loop DBS is an emerging neuromodulation pattern in Parkinson's disease with dyanmic adjustment of stimulation parameters to patients' disease fluctuations and state of activity. The purpose of this study is to verify the long-term safety and effectiveness of closed-loop DBS. Through comparing with open-loop DBS, the study also determine whether closed-loop DBS is more effective than conventional open-loop DBS on PD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary Parkinson's disease: Diagnosis of primary Parkinson's disease should meet the diagnostic criteria outlined in the "Diagnosis Standards for Parkinson's Disease in China" published in 2016 or the diagnostic criteria for primary Parkinson's disease by the International Parkinson and Movement Disorder Society (MDS) published in 2015.
2. Good response to levodopa combination therapy.
3. Significant reduction in drug efficacy or significant impact on the patient's quality of life due to prominent motor complications.
4. Intolerable adverse reactions to medication affecting its efficacy.
5. Presence of uncontrollable tremors despite medication.

Exclusion Criteria:

1. Patients who have undergone pallidotomy or other brain surgeries.
2. Patients with secondary Parkinson syndromes or Parkinson plus syndromes.
3. Patients with concurrent central nervous system and peripheral nervous system diseases.
4. Patients with severe systemic diseases, unstable vital signs, or those who cannot tolerate clinical assessments.
5. Patients with severe psychiatric disorders.
6. Patients who are unable to provide informed consent due to cognitive or communication impairments or those who refuse to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Movement disorders evaluation | 1-3 days
  Using MDS-UPDRS III rating scale （0-132, the higher score means a worse outcome） and Rush dyskinesia rating scale （0-12, the higher score means a worse outcome） combined with IMU to evaluate the motor function improvement under both closed-loop DBS and open-loop DBS condition
Sleep Structure Evaluation | 1-3 nights
  Using polysomnography evaluation （sleep efficiency，N1/N2/N3/REM/Wake after sleep onset duration and percentage，arousal index） and subjuective sleep quality rating scale to evaluate the sleep improvement under both closed-loop DBS and open-loop DBS condition
Diary Outcomes in Parkinson's Disease | 1-3days
  Using SCOPA-DC （0-87, the higher score means a worse outcome） to evaluate the diary outcomes under both closed-loop DBS and open-loop DBS condition

SECONDARY OUTCOMES:
Safety (Stimulation-related AEs) and Subjective Satisfactory | 1-3days
  Number of modulation related Adverse Events or abnormal vital signs.
Total Electrical Energy Delivered to patients | 1-3days
  To evaluate the energy changes in closed-loop DBS and open-loop DBS modualtion

OTHER OUTCOMES:
Neurophysiological changes of STN-LFP in daytime and sleep | at 3,6,9,12,15 months compared to baseline
  Changes of the power and entropy features of delta, theta, alpha, beta and gamma oscillations
Functional connectivity changes during long-term DBS modulation | at 3,6,9,12,15 months compared to baseline
  Changes of subcortical and cortical functional connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- National Engineering Research Center of Neuromodulation, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No